CLINICAL TRIAL: NCT04808297
Title: A Study in Subjects With Neuronal Ceroid Lipofuscinoses Taking Trehalose
Brief Title: Trehalose in Subjects With Neuronal Ceroid Lipofuscinoses
Acronym: 3AL-CLN36
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Filippo Maria Santorelli, Director Molecular Medicine, Neurogenetics and Neuromuscular Disorders, IRCCS Fondazione Stella Maris
Other Study IDs: 3AL-CLN36
Record Dates: First submitted 2021-03-02; First posted 2021-03-22 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Neuronal Ceroid-Lipofuscinoses
Keywords: Juvenile Neuronal Ceroid-Lipofuscinoses; Unified Batten Disease Rating Scale
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuronal Ceroid Lipofuscinoses (NCL) or Batten's disease are the most common juvenile neurodegenerative disease, characterized by early blindness, movement disorders, cognitive and behavioral impairment, epilepsy, and retinopathy.

This study aims to collect clinical and laboratory data of patients with NCL taking Trehalose.

DETAILED DESCRIPTION:
This study aims to collect clinical and laboratory data of patients with NCL taking Trehalose.

ELIGIBILITY:
Inclusion Criteria:

* NCL genetic diagnosis (mutation in genes CLN3 or CLN6)
* Signed informed consent

Exclusion Criteria:

* Other concomitant neurodegenerative diseases.
* Therapeutic and eating changes in the last four months prior to the study
* Unstable clinical conditions (myoclonus worsening, instability in sleep, parenteral nutrition)
* Refusal to sign the informed consent

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects in regular clinical practice affected by CLN3 o CLN6 diagnose by genetic tests
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline clinical status assessed using Annex VII of the Unified Batten Disease Rating Scale (UBDRS) (score 0-5 where 5 is the worst outcome) at 12 and 24 months | month 0, month 12, month 24
  Blood samples

SECONDARY OUTCOMES:
Change from Baseline using Annex VII of Unified Batten Disease Rating Scale (UBDRS) (score 0-5 where 5 is the worst outcome) at 12 and 24 months | month 0, month 12, month 24
  Blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajaj L, Lotfi P, Pal R, Ronza AD, Sharma J, Sardiello M. Lysosome biogenesis in health and disease. J Neurochem. 2019 Mar;148(5):573-589. doi: 10.1111/jnc.14564. Epub 2018 Oct 18. PMID 30092616
- [Background] Lee HJ, Yoon YS, Lee SJ. Mechanism of neuroprotection by trehalose: controversy surrounding autophagy induction. Cell Death Dis. 2018 Jun 15;9(7):712. doi: 10.1038/s41419-018-0749-9. PMID 29907758
- [Background] Palmieri M, Pal R, Nelvagal HR, Lotfi P, Stinnett GR, Seymour ML, Chaudhury A, Bajaj L, Bondar VV, Bremner L, Saleem U, Tse DY, Sanagasetti D, Wu SM, Neilson JR, Pereira FA, Pautler RG, Rodney GG, Cooper JD, Sardiello M. mTORC1-independent TFEB activation via Akt inhibition promotes cellular clearance in neurodegenerative storage diseases. Nat Commun. 2017 Feb 6;8:14338. doi: 10.1038/ncomms14338. PMID 28165011
- [Background] Sardiello M. Transcription factor EB: from master coordinator of lysosomal pathways to candidate therapeutic target in degenerative storage diseases. Ann N Y Acad Sci. 2016 May;1371(1):3-14. doi: 10.1111/nyas.13131. PMID 27299292
- [Background] Schulz A, Ajayi T, Specchio N, de Los Reyes E, Gissen P, Ballon D, Dyke JP, Cahan H, Slasor P, Jacoby D, Kohlschutter A; CLN2 Study Group. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med. 2018 May 17;378(20):1898-1907. doi: 10.1056/NEJMoa1712649. Epub 2018 Apr 24. PMID 29688815